CLINICAL TRIAL: NCT01074463
Title: A Relative Bioavailability Study of 0.25 mg Pramipexole Dihydrochloride Tablets Under Non-Fasting Conditions
Brief Title: Pramipexole Dihydrochloride 0.25 mg Tablets Under Non-Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: R04-1203
Record Dates: First submitted 2010-02-22; First posted 2010-02-24 (Estimated); Results first posted 2010-04-30 (Estimated); Last update posted 2010-04-30 (Estimated); Status verified 2010-04

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Pramipexole

ARMS (2):
- 1 (Experimental): Pramipexole Dihydrochloride 0.25 mg Tablets
  Interventions: Drug: Pramipexole Dihydrochloride
- 2 (Active Comparator): Mirapex® 0.25 mg Tablets
  Interventions: Drug: Pramipexole Dihydrochloride

INTERVENTIONS:
Drug: Pramipexole Dihydrochloride — 0.25 mg Tablet
  Arms: 1
Drug: Pramipexole Dihydrochloride — 0.25 mg Tablet
  Other Names: Mirapex®
  Arms: 2

SUMMARY:
The object of this study was to compare the relative bioavailability (rate and extent of absorption) of Pramipexole Dihydrochloride Tablets 0.25 mg by Barr Laboratories, Inc. with that of Mirapex® Tablets 0.25 mg distributed by Boehringer Ingelheim Pharmaceuticals, Inc. following a single oral dose in healthy adults under non-fasting conditions.

DETAILED DESCRIPTION:
Criteria for Evaluation: FDA Bioequivalence Criteria

Statistical Methods: FDA Bioequivalence Statistical Methods

ELIGIBILITY:
Inclusion Criteria:

* All volunteers selected for this study will be healthy men and women 18 to 45 years of age, inclusive.
* The weight range will not exceed + 20% for height and body frame as per "Desirable Weights for Adults - 1983 Metropolitan Height and Weight Table"
* Each volunteer will complete the screening process within 28 days prior to Period 1 dosing.
* Consent documents for both the screening evaluation and HIV antibody determination will be reviewed, discussed, and signed by each potential participant before full implementation of screening procedures.
* If female: and of child bearing potential is practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), is postmenopausal for at least 1 year, or is surgically sterile.

Exclusion Criteria:

* Volunteers with a recent history of drug or alcohol addiction or abuse.
* Volunteers with the presence of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurologic system(s) or psychiatric disease (as determined by the clinical investigator).
* Volunteers whose clinical laboratory test values are outside the accepted reference range and when confirmed on re-examination are deemed to be clinically significant.
* Volunteers demonstrating a reactive screen for hepatitis B surface antigen, hepatitis C antibody, or HIV antibody.
* Volunteers demonstrating a positive drug abuse screen when screened for this study.
* Female volunteers demonstrating a positive pregnancy screen.
* Female volunteers who are currently breastfeeding.
* Volunteers with a history of allergic response(s) to pramipexole or related drugs.
* Volunteers with a history of clinically significant allergies including drug allergies.
* Volunteers with a clinically significant illness during the 4 weeks prior to Period I dosing (as determined by the clinical investigators).
* Volunteers who currently use tobacco products.
* Volunteers who have taken any drug known to induce or inhibit hepatic drug metabolism in the 28 days prior to Period I dosing.
* Volunteers who report donating greater than 150 mL of blood within 28 days prior to Period I dosing. All subjects will be advised not to donate blood for 4 weeks after completing the study.
* Volunteers who have donated plasma (e.g. plasmapheresis) within 14 days prior to Period I dosing. All subjects will be advised not to donate plasma for 4 weeks after completing the study.
* Volunteers who report receiving any investigational drug within 28 days prior to Period I dosing.
* Volunteer who report taking any systemic prescription medication in the 14 days prior to Period I dosing. Diltiazem (Cardizem®), triamterene (Dyrenium®), verapamil (Calan®, Covera-HS®), quinidine, and quinine are prohibited throughout the entire study.
* Volunteers using OTC medication 7 days prior to dosing including vitamins, cough and cold preparations. Cimetidine (Tagamet®), ranitidine (Zantac®), probenecid (Pro-Bionate®), and any OTC antihistamine products (such as diphenhydramine, chlorpheniramine) are absolutely prohibited throughout the entire study.
* Volunteers who consume food containing poppy seeds in the 48 hours before dosing of each period.
* Volunteers who consume grapefruit or related products 14 days prior to Period I dosing.
* Female volunteers who report the use of oral contraceptives or injectable contraceptives.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2005-02; Primary Completion 2005-03 (Actual); Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D Carlson, Pharm. D, Principal Investigator — PRACS Institute, Ltd.
Locations (1):
- PRACS Institute, Ltd., Fargo, North Dakota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Test (Pramipexole Dihydrochloride) First: 0.25 mg Pramipexole Dihydrochloride Tablets test product dosed in first period followed by 0.25 mg Mirapex® Tablets reference product dosed in the second period.
- Reference (Mirapex®) First: 0.25 mg Mirapex® Tablets reference product dosed in first period followed by 0.25 mg Pramipexole Dihydrochloride Tablets test product dosed in the second period.
Period: First Intervention
Arm/Group | Test (Pramipexole Dihydrochloride) First | Reference (Mirapex®) First
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Washout of 7 Days
Arm/Group | Test (Pramipexole Dihydrochloride) First | Reference (Mirapex®) First
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Test (Pramipexole Dihydrochloride) First | Reference (Mirapex®) First
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Test (Pramipexole Dihydrochloride) First | Reference (Mirapex®) First | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 12 | 24
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 7 | 12
  Male | 7 | 5 | 12
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 10 | 12 | 22
  Black | 1 | 0 | 1
  Native American | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Cmax (Maximum Observed Concentration of Drug Substance in Plasma)
Description: Bioequivalence based on Cmax.
Time Frame: Blood samples collected over a 48 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Test (Pramipexole Dihydrochloride): 0.25 mg Pramipexole Dihydrochloride Tablets test product dosed in either period.
- Reference (Mirapex®): 0.25 mg Mirapex® Tablets reference product dosed in either period.
Arm/Group | Test (Pramipexole Dihydrochloride) | Reference (Mirapex®)
Number analyzed (Participants) | 24 | 24
ng/mL | 0.61 (0.22) | 0.54 (0.10)
Statistical Analysis 1: Comparison: Test (Pramipexole Dihydrochloride) vs Reference (Mirapex®); Test type: Non-Inferiority or Equivalence — The ANOVA model was utilized in comparing the effects between the test and reference products. Differences were declared statistically significant at the 5% level (p<0.05); Ratio of the T/R geometric mean x 100 = 109.18, 90% CI 2-sided [99.25 to 120.12] — Bioequivalence is established if the 90% confidence interval for the ln-transformed geometric mean between the reference and test product fall within the interval of 80-125%

2. Primary Outcome: AUC0-t (Area Under the Concentration-time Curve From Time Zero to Time of Last Measurable Concentration)
Description: Bioequivalence based on AUC0-t.
Time Frame: Blood samples collected over a 48 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Test (Pramipexole Dihydrochloride) | Reference (Mirapex®)
Number analyzed (Participants) | 24 | 24
ng*h/mL | 5.86 (1.18) | 5.68 (1.36)
Statistical Analysis 1: Comparison: Test (Pramipexole Dihydrochloride) vs Reference (Mirapex®); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 104.06, 90% CI 2-sided [98.73 to 109.68] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: AUC0-inf (Area Under the Concentration-time Curve From Time Zero to Infinity)
Description: Bioequivalence based on AUC0-inf.
Time Frame: Blood samples collected over a 48 hour period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Test (Pramipexole Dihydrochloride) | Reference (Mirapex®)
Number analyzed (Participants) | 24 | 24
ng*h/mL | 6.27 (1.21) | 6.17 (1.40)
Statistical Analysis 1: Comparison: Test (Pramipexole Dihydrochloride) vs Reference (Mirapex®); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 102.34, 90% CI 2-sided [97.78 to 107.11] — [estimate comment as in outcome 1, analysis 1]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the course of the study, which was approximately 2 weeks in duration.
Description: Volunteers were monitored throughout the study for any adverse experiences. AEs were collected through both solicited and unsolicited methods. The volunteers were encouraged to report signs, symptoms, and any changes in health to the clinic staff.
Arm/Group | Test (Pramipexole Dihydrochloride) First | Reference (Mirapex®) First
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 2/24 | 4/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Test (Pramipexole Dihydrochloride) First (N=24) | Reference (Mirapex®) First (N=24)
Dizziness (General disorders) | 2 (2) | 0 (0)
Headache (General disorders) | 0 (0) | 2 (2)
Nausea (General disorders) | 0 (0) | 2 (2)
Nervousness (General disorders) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator is not permitted to discuss or publish trial results.